CLINICAL TRIAL: NCT02425501
Title: Special Drug Use Investigation of EYLEA for Diabetic Macular Edema
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17544; EY1510JP (Other: Company internal)
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Macular Edema
Keywords: Aflibercept; anti-VEGF
MeSH Terms: conditions — Macular Edema | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aflibercept (Eylea,BAY86-5321): Decision of EYLEA treatment is made by attending investigator according to the Japanese Package Insert
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY86-5321) — Administration by intravitreal injection

SUMMARY:
The objectives of this study are to investigate the safety and effectiveness of EYLEA

DETAILED DESCRIPTION:
This is a prospective, non-interventional, multi center post-authorization safety study that includes patients with a diagnosis of myopic choroidal neovascularization. The investigator will have made the choice of treatment (EYLEA) as well as the decision to use EYLEA according the Japanese Package Insert prior to enrolling the patient in this study.

The observation period for each patient starts when therapy with EYLEA is initiated. The enrollment period is 2 years. Patients will be followed for a time period of 2 years or until it is no longer possible (e.g. lost to follow-up) within the 2 years. In total, 600 patients will be recruited.

For each patient, data are collected as defined in the electronic case report form (eCRF) at the initial visit, follow-up visits and final visit, either by routine clinical visits (as per investigators routine practice).

ELIGIBILITY:
Inclusion Criteria:

* Patients who start EYLEA treatment for Diabetic Macular Edema (DME)

Exclusion Criteria:

* Patients who have already received EYLEA treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female and male patients with DME diagnosis will be enrolled after the investigators have taken the decision for the treatment with EYLEA. Those patients who have had EYLEA prescribed previously will not be included in this study. Physicians should consult the full prescribing information for EYLEA before enrolling patients and be familiarized with the safety information in the product package label.
Sampling Method: Non-Probability Sample
Enrollment: 646 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Number of participants of Adverse Events | Up to 12 months
Number of participants of Serious Adverse Events | Up to 12 months

SECONDARY OUTCOMES:
Mean change in visual acuity from baseline to 12 months | Baseline to 12 months
Mean change in retina thickness from baseline to 12 months | Baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Derived] Sugimoto M, Handa C, Hirano K, Sunaya T, Kondo M. Intravitreal aflibercept for diabetic macular edema in real-world clinical practice in Japan: 24-month outcomes. Graefes Arch Clin Exp Ophthalmol. 2022 Nov;260(11):3489-3498. doi: 10.1007/s00417-022-05703-9. Epub 2022 Jun 2. PMID 35652946
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/